CLINICAL TRIAL: NCT02004275
Title: A Phase I/II Study of Pomalidomide, Dexamethasone and Ixazomib vs. Pomalidomide and Dexamethasone for Patients With Multiple Myeloma Relapsing on Lenalidomide as Part of First Line Therapy
Brief Title: Pomalidomide and Dexamethasone With or Without Ixazomib in Treating Patients With Relapsed Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Celgene Corporation (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A061202; NCI-2013-01702 (Registry Identifier: Clinical Trial Reporting Program); U10CA031946 (NIH)
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma in Relapse
MeSH Terms: interventions — pomalidomide; ixazomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (pomalidomide, dexamethasone) (Experimental): Patients receive pomalidomide PO QD on days 1-21 and dexamethasone PO QD on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving disease progression may cross over to Arm II.
  Interventions: Drug: pomalidomide; Drug: dexamethasone
- Arm II (pomalidomide, dexamethasone, ixazomib) (Experimental): Patients receive pomalidomide, dexamethasone, and ixazomib as in Phase I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pomalidomide; Drug: ixazomib; Drug: dexamethasone

INTERVENTIONS:
Drug: pomalidomide — given PO
  Other Names: Pomalyst®
Drug: ixazomib — given PO
  Other Names: MLN9708
  Arms: Arm II (pomalidomide, dexamethasone, ixazomib)
Drug: dexamethasone — given PO

SUMMARY:
This randomized phase I/II trial studies the side effects and best dose of pomalidomide and ixazomib when given together with dexamethasone and to see how well pomalidomide and dexamethasone with or without ixazomib works in treating patients with multiple myeloma that has come back. Biological therapies, such as pomalidomide and dexamethasone, may stimulate the immune system in different ways and stop cancer cells from growing. Ixazomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It is not yet known whether pomalidomide and dexamethasone are more effective with or without ixazomib in treating multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) for combination therapy pomalidomide/dexamethasone/ixazomib. (Phase I) II. To assess whether the combination of pomalidomide/dexamethasone/ixazomib improves progression-free survival (PFS) relative to pomalidomide/dexamethasone. (Phase II)

SECONDARY OBJECTIVES:

I. To determine dose-limiting toxicities (DLTs). (Phase I) II. To analyze type and grade of all serious adverse events (SAEs). (Phase I) III. To analyze type and grade of all adverse events (AEs). (Phase I) IV. To analyze the reason for and incidence of dose modifications/omissions/delays. (Phase I) V. To assess preliminary evidence of clinical efficacy. (Phase I) VI. To assess whether the overall response rate (ORR), partial response (PR), very good partial response (VGPR), complete response (CR) or stringent CR (sCR) rate differ with respect to treatment regimen. (Phase II) VII. To assess the clinical benefit rate (CBR: minimal response [MR] + ORR) for pomalidomide/dexamethasone/ixazomib compared to pomalidomide/dexamethasone. (Phase II) VIII. To assess the disease control rate (DCR: stable disease [SD] + CBR) for pomalidomide/dexamethasone/ixazomib compared to pomalidomide/dexamethasone. (Phase II) IX. For those patients achieving a PR or better, we will assess whether the combination of pomalidomide/dexamethasone/ixazomib increases the duration of response (DOR) compared to pomalidomide/dexamethasone. (Phase II) X. To assess whether the combination of pomalidomide/dexamethasone/ixazomib improves overall survival (OS) compared to those taking pomalidomide/dexamethasone alone. (Phase II) XI. To assess time to next treatment (TNT) for patients taking pomalidomide/dexamethasone/ixazomib compared to those on pomalidomide/dexamethasone. (Phase II) XII. To evaluate the safety of pomalidomide/dexamethasone/ixazomib compared with pomalidomide/dexamethasone. (Phase II) XIII. For patients on the pomalidomide/dexamethasone arm who opt to cross-over to the pomalidomide/dexamethasone/ixazomib arm, assessment of response rate (ORR, CBR, DCR), DOR, TNT, PFS and OS will be evaluated from date of cross-over. (Phase II) XIV. To determine if baseline level of perceived fatigue and overall quality of life (QOL) is associated with OS. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of pomalidomide and ixazomib followed by a phase II study.

After completion of study treatment, patients are followed up every 4 weeks until disease progression and then every 3 months for 3 years.

ELIGIBILITY:
* Histologically confirmed diagnosis of symptomatic multiple myeloma; relapsed disease is myeloma that has previously responded to prior therapy (MR or better) and subsequently progressed
* Patient must have measurable disease or non-measurable disease, defined as one or more of the following holding true:

  * Measurable disease:

    * Serum M-protein >= 1.0 g/dL (>= 0.5 g/dL for IgA or IgM myeloma) and/or
    * Urine M-protein >= 200 mg/24 hours and/or
    * Involved serum free light chain level >= 10 mg/dL AND an abnormal serum free light chain ratio
  * For non-measurable disease:

    * Baseline marrow burden of myeloma of at least 30%
* Progression on lenalidomide as part of first line therapy (lenalidomide-refractory disease)

  * Lenalidomide-refractory disease is defined as disease progression on or progression within 60 days of the last dose of a lenalidomide-based treatment; patients should have received at least 2 cycles of a lenalidomide-based regimen to be evaluable for refractoriness; examples: 1) progression on lenalidomide maintenance therapy after initial induction +/- consolidation; 2) initial response followed by progression on continuous lenalidomide-dexamethasone +/- elotuzumab or daratumumab
* Pomalidomide naive disease
* Proteasome inhibitor naive or sensitive disease; proteasome inhibitor sensitive disease is defined as a PR or better to prior proteasome inhibitor-based therapy that is maintained for >= 60 days from the last dose of the proteasome inhibitor

  * A patient who receives induction therapy with lenalidomide, bortezomib and dexamethasone and achieves a PR or better but subsequently progresses on continued lenalidomide or lenalidomide-dexamethasone would be eligible provided the progression occurs 60 days or more after discontinuation of the bortezomib; similarly, ixazomib exposure is allowed provided they meet the definition of proteasome inhibitor sensitive disease
* 1 prior line of systemic therapy for multiple myeloma, where a line of therapy for myeloma is defined as 1 or more planned cycles of single agent or combination therapy, as well as a planned series of treatment regimens administered in a sequential manner (e.g. lenalidomide, bortezomib and dexamethasone induction therapy for 4 cycles followed by autologous stem cell transplantation and then lenalidomide maintenance therapy would be considered 1 line of prior therapy); a new line of therapy begins when a planned therapy is modified to include other treatment agents (alone or in combination) as a result of disease progression, disease relapse or treatment-related toxicity (e.g. a patient is progressing in the face of lenalidomide maintenance therapy and has bortezomib and dexamethasone added into their regimen); a new line of therapy also begins when a planned treatment-free interval is interrupted by the need to start treatment due to disease relapse/progression (e.g. a patient with relapsed myeloma achieves a partial response after a planned 8 cycles of cyclophosphamide, bortezomib and dexamethasone, enjoys an 8-month period off therapy but then experiences disease progression requiring re-initiation of therapy)
* Allogeneic stem cell transplantation is allowed provided the patient is >= 1 year from transplant at time of registration, is not on immunosuppressive therapy to treat/prevent graft-versus-host disease, has no evidence of active graft versus host disease, and no evidence of active infection
* No other chemotherapy or radiation therapy within 14 days prior to registration
* No investigational therapy within 14 days prior to registration
* No major surgery within 28 days prior to registration
* No G-CSF (filgrastim) or GM-CSF (sargramostim) within 7 days of registration or pegfilgrastim within 14 days of registration to meet eligibility criteria
* No platelet transfusions within 7 days of registration to meet eligibility criteria; Note: red blood cell transfusions are allowed at any time
* A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)

  * Women of childbearing potential:

    * Must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mlU/ml no more than 14 days prior to registration and must agree to repeat this test within 24 hours of starting pomalidomide
    * Must either commit to complete abstinence from heterosexual contact or begin TWO acceptable methods of birth control, one highly effective method and one additional effective (barrier) method, AT THE SAME TIME, before starting pomalidomide
    * Must agree to ongoing pregnancy testing
    * Must agree to not become pregnant or breast feed a child during treatment on this protocol
  * Men must practice complete abstinence or agree to use a condom during sexual contact with a female of childbearing potential, even if they have had a successful vasectomy
  * Note: All participants must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Platelet count >= 50 x 10^9/L
* Calculated (Calc.) creatinine clearance >= 30 mL/min; calculated utilizing the Cockcroft-Gault formula or 24-hour urine collection
* Total bilirubin < 1.5 x upper limits of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x upper limits of normal (ULN)
* Note: G-CSF and platelet transfusions cannot be used to increase counts to meet eligibility criteria
* Patients cannot have:

  * Central nerve system involvement
  * Primary refractory multiple myeloma, where primary refractory multiple myeloma is defined as disease that is nonresponsive - patients who have never achieved a minimal response (MR) or better - with any therapy over the course of their disease; it includes patients who never achieve MR or better in whom there is no significant change in M-protein and no evidence of clinical progression as well as patients who meet criteria for true progressive disease (PD)
  * Primary or secondary plasma cell leukemia
  * Light-chain (AL) amyloidosis or polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome
  * Known active hepatitis C based on:

    * +hepatitis C virus (HCV) antibody (confirmed)
    * +HCV RNA
    * Liver disease with history of positive serology
    * Note: patients with a prior history of hepatitis C that has been successfully eradicated with antiviral therapy are eligible
  * Known hepatitis B surface antigen positivity
  * Previous hypersensitivity to any of the components of the study treatment
  * Prior history of erythema multiforme with thalidomide or lenalidomide treatment
* =< grade 2 peripheral neuropathy
* Adequate cardiac function, defined as:

  * No electrocardiogram (EKG) evidence of acute ischemia
  * No EKG evidence of active, clinically significant conduction system abnormalities
  * No EKG evidence of > grade 2 (> 480 ms) corrected QT (QTc) prolongation
  * Prior to study entry, any EKG abnormality at screening not felt to put the patient at risk has to be documented by the investigator as not medically significant
  * No uncontrolled angina or severe ventricular arrhythmias
  * No clinically significant pericardial disease
  * No history of myocardial infarction within 6 months prior to registration
  * No class 3 or higher New York Heart Association congestive heart failure
* No strong inducers of cytochrome P450 (CYP) 3A4 or CYP1A2 or strong inhibitors of CYP3A4 or CYP1A2 within 14 days prior to registration

  * Note: Ixazomib is a substrate of CYP3A4 and CYP1A2
* Patients with human immunodeficiency virus (HIV) infection are eligible, provided they meet the following:

  * No history of acquired immunodeficiency syndrome (AIDS)-defining conditions or other HIV related illness
  * Cluster of differentiation (CD)4+ cells nadirs > 350/mm^3 within 28 days prior to registration
  * Treatment sensitive HIV and, if on anti-HIV therapy, HIV viral load < 50 copies/mm^3 within 28 days prior to registration
  * Note: HIV+ patients who enroll on this study and are assigned to treatment with ixazomib may need to modify their anti-retroviral therapy prior to receiving protocol therapy if they are on strong inducers or potent inhibitors of cytochrome P450 3A4
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): Patients randomized to Arm 1 may opt to switch to the 3-drug regimen following disease progression; these patients must be re-registered to the study and meet the eligibility criteria below
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): Patient must have measurable disease or non-measurable disease after progression on pomalidomide + dexamethasone, defined as one or more of the following holding true:

  * Measurable disease:
  * Serum M-protein >= 0.5 g/dL and/or
  * Urine M-protein >= 200 mg/24 hours and/or
  * Involved serum free light chain level >= 10 mg/dL AND an abnormal serum free light chain ratio

    * For non-measurable disease:
  * Marrow burden of myeloma of at least 30%
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2):

  * Women of childbearing potential:

    ** Must have a negative serum or urine pregnancy test within 72 hours prior to re-registration

    ** Must either commit to complete abstinence from heterosexual contact or begin TWO acceptable methods of birth control, one highly effective method and one additional effective (barrier) method, AT THE SAME TIME, before starting pomalidomide

    ** Must agree to ongoing pregnancy testing

    ** Must agree to not become pregnant or breast feed a child during treatment on this protocol
  * Men must practice complete abstinence or agree to use a condom during sexual contact with a female of childbearing potential, even if they have had a successful vasectomy
  * Note: All participants must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): ECOG performance status 0-2
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): Platelet count >= 50 x 10^9/L
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): Calc. creatinine clearance >= 30 mL/min

  * Calculated utilizing the Cockcroft-Gault formula or 24-hour urine collection
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): Total bilirubin < 1.5 x upper limits of normal (ULN)
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): AST and ALT < 2.5 x upper limits of normal (ULN)
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): Note: G-CSF and platelet transfusions cannot be used to increase counts to meet eligibility criteria
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): =< grade 2 peripheral neuropathy
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): No strong inducers of cytochrome P450 (CYP) 3A4 or CYP1A2 or strong inhibitors of CYP3A4 or CYP1A2 * Note: Ixazomib is a substrate of CYP3A4 and CYP1A2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Voorhees, MD, Study Chair — University of North Carolina, Chapel Hill
Locations (336):
- United States (336):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Rex Hematology Oncology Associates-Blue Ridge, Raleigh, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Voorhees P, Suman V, Efebera Y, Raje N, Tuchman S, Rodriguez C, Laubach J, Bova-Solem M, Carlisle D, Usmani S, McCarthy P, Richardson PG. Alliance A061202: ixazomib, pomalidomide, and dexamethasone for patients with lenalidomide-refractory MM in first relapse. Blood Adv. 2024 Oct 8;8(19):5039-5050. doi: 10.1182/bloodadvances.2024013623. PMID 39058954
- [Derived] Voorhees PM, Suman VJ, Tuchman SA, Laubach JP, Hassoun H, Efebera YA, Mulkey F, Bova-Solem M, Santo K, Carlisle D, McCarthy PL, Richardson PG. A phase I/II study of ixazomib, pomalidomide, and dexamethasone for lenalidomide and proteasome inhibitor refractory multiple myeloma (Alliance A061202). Am J Hematol. 2021 Dec 1;96(12):1595-1603. doi: 10.1002/ajh.26361. Epub 2021 Oct 6. PMID 34559902

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Pomalidomide, Dexamethasone): Patients receive 4mg of pomalidomide PO QD on days 1-21 and 40mg dexamethasone PO QD on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving disease progression may cross over to Arm II.
- Arm II (Pomalidomide, Dexamethasone, Ixazomib): Patients receive 4mg pomalidomide, 40mg dexamethasone, and 4mg ixazomib as in Phase I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 1: A 3 + 3 phase I dose escalation design was used to examine the safety profile and establish the MTD of IXA when given in combination with POM-DEX. Protocol therapy was administered over a 28-day cycle. IXA was given at a dose of 2.3 up to 4 mg by mouth on days 1, 8, and 15; POM at 2 up to 4 mg daily by mouth on days 1-21; and DEX 20 mg (age > 75 years) or 40 mg (age ≤ 75) by mouth on days 1, 8, 15, and 22 (Table 1). A new cycle of treatment was not to begin until the ANC was ≥ 1.0 × 109/L, platelets ≥ 50 × 109/L, and all other adverse events (AEs) had improved to grade 1 or baseline. Treatment continued until PD, the emergence of unacceptable toxicity, or patient request to discontinue protocol treatment. Dose Level 1 was 2mg POM-DEX and 3mg IXA.
- Phase I Dose Level 2: A 3 + 3 phase I dose escalation design was used to examine the safety profile and establish the MTD of IXA when given in combination with POM-DEX. Protocol therapy was administered over a 28-day cycle. IXA was given at a dose of 2.3 up to 4 mg by mouth on days 1, 8, and 15; POM at 2 up to 4 mg daily by mouth on days 1-21; and DEX 20 mg (age > 75 years) or 40 mg (age ≤ 75) by mouth on days 1, 8, 15, and 22 (Table 1). A new cycle of treatment was not to begin until the ANC was ≥ 1.0 × 109/L, platelets ≥ 50 × 109/L, and all other adverse events (AEs) had improved to grade 1 or baseline. Treatment continued until PD, the emergence of unacceptable toxicity, or patient request to discontinue protocol treatment. Dose Level 2 was 3mg POM-DEX and 3mg IXA.
- Phase 1 Dose Level 3: A 3 + 3 phase I dose escalation design was used to examine the safety profile and establish the MTD of IXA when given in combination with POM-DEX. Protocol therapy was administered over a 28-day cycle. IXA was given at a dose of 2.3 up to 4 mg by mouth on days 1, 8, and 15; POM at 2 up to 4 mg daily by mouth on days 1-21; and DEX 20 mg (age > 75 years) or 40 mg (age ≤ 75) by mouth on days 1, 8, 15, and 22 (Table 1). A new cycle of treatment was not to begin until the ANC was ≥ 1.0 × 109/L, platelets ≥ 50 × 109/L, and all other adverse events (AEs) had improved to grade 1 or baseline. Treatment continued until PD, the emergence of unacceptable toxicity, or patient request to discontinue protocol treatment. Dose Level 3 was 4mg POM-DEX and 3mg IXA.
- Phase 1 Dose Level 4: A 3 + 3 phase I dose escalation design was used to examine the safety profile and establish the MTD of IXA when given in combination with POM-DEX. Protocol therapy was administered over a 28-day cycle. IXA was given at a dose of 2.3 up to 4 mg by mouth on days 1, 8, and 15; POM at 2 up to 4 mg daily by mouth on days 1-21; and DEX 20 mg (age > 75 years) or 40 mg (age ≤ 75) by mouth on days 1, 8, 15, and 22 (Table 1). A new cycle of treatment was not to begin until the ANC was ≥ 1.0 × 109/L, platelets ≥ 50 × 109/L, and all other adverse events (AEs) had improved to grade 1 or baseline. Treatment continued until PD, the emergence of unacceptable toxicity, or patient request to discontinue protocol treatment. Dose Level 4 was 4mg POM-DEX and 4mg IXA.
Period: Phase 1
Arm/Group | Arm I (Pomalidomide, Dexamethasone) | Arm II (Pomalidomide, Dexamethasone, Ixazomib) | Phase 1 Dose Level 1 | Phase I Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4
Started | 0 | 0 | 3 | 5 | 7 | 11
Completed | 0 | 0 | 3 | 3 | 6 | 6
Not Completed | 0 | 0 | 0 | 2 | 1 | 5
Not completed — Ineligible | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 5
Period: Phase 2 Part 1
Arm/Group | Arm I (Pomalidomide, Dexamethasone) | Arm II (Pomalidomide, Dexamethasone, Ixazomib) | Phase 1 Dose Level 1 | Phase I Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4
Started | 45 | 47 | 0 | 0 | 0 | 0
Completed | 39 | 38 | 0 | 0 | 0 | 0
Not Completed | 6 | 9 | 0 | 0 | 0 | 0
Not completed — Ineligible | 6 | 9 | 0 | 0 | 0 | 0
Period: Phase 2 Part 2
Arm/Group | Arm I (Pomalidomide, Dexamethasone) | Arm II (Pomalidomide, Dexamethasone, Ixazomib) | Phase 1 Dose Level 1 | Phase I Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4
Started | 30 | 0 | 0 | 0 | 0 | 0
Completed | 26 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase II Arm I (Pomalidomide, Dexamethasone): Patients receive pomalidomide PO QD on days 1-21 and dexamethasone PO QD on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving disease progression may cross over to Arm II.
- Phase II Arm II (Pomalidomide, Dexamethasone, Ixazomib): Patients receive pomalidomide, dexamethasone, and ixazomib as in Phase I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 2: A 3 + 3 phase I dose escalation design was used to examine the safety profile and establish the MTD of IXA when given in combination with POM-DEX. Protocol therapy was administered over a 28-day cycle. IXA was given at a dose of 2.3 up to 4 mg by mouth on days 1, 8, and 15; POM at 2 up to 4 mg daily by mouth on days 1-21; and DEX 20 mg (age > 75 years) or 40 mg (age ≤ 75) by mouth on days 1, 8, 15, and 22 (Table 1). A new cycle of treatment was not to begin until the ANC was ≥ 1.0 × 109/L, platelets ≥ 50 × 109/L, and all other adverse events (AEs) had improved to grade 1 or baseline. Treatment continued until PD, the emergence of unacceptable toxicity, or patient request to discontinue protocol treatment. Dose Level 2 was 3mg POM-DEX and 3mg IXA.
- Total: Total of all reporting groups
Arm/Group | Phase II Arm I (Pomalidomide, Dexamethasone) | Phase II Arm II (Pomalidomide, Dexamethasone, Ixazomib) | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4 | Total
Number analyzed (Participants) | 45 | 47 | 3 | 5 | 7 | 11 | 118
Age, Continuous [Median (Full Range); unit: years] | 65 [41 to 85] | 67 [41 to 83] | 64.0 [57 to 72] | 63 [47 to 77] | 65 [59 to 69] | 69 [51 to 80] | 66 [41 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 25 | 1 | 1 | 4 | 4 | 52
  Male | 28 | 22 | 2 | 4 | 3 | 7 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 0 | 1 | 0 | 2 | 8
  Not Hispanic or Latino | 33 | 43 | 3 | 3 | 6 | 9 | 97
  Unknown or Not Reported | 8 | 3 | 0 | 1 | 1 | 0 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 6 | 1 | 0 | 1 | 0 | 13
  White | 37 | 39 | 2 | 5 | 6 | 8 | 97
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 0 | 0 | 0 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Pomalidomide and Ixazomib, Determined According to Incidence of Dose Limiting Toxicity (DLT) Graded Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (Phase I)
Description: For this protocol, dose-limiting toxicity (DLT) will be defined by the following adverse events at least possibly related to study therapy: Grade 3 or higher non-hematologic toxicity, with the following exceptions: Alopecia is not expected but would not be considered a DLT. Nausea, vomiting and diarrhea will only be considered a DLT if it cannot be adequately managed with optimal supportive care. Grade 3 or 4 hyperglycemia due to dexamethasone will only be considered a DLT if it cannot be controlled with appropriate therapy Grade 4 hematologic toxicity, with the following exceptions: Grade 4 lymphopenia is expected with this regimen and will not be construed as a DLT. Grade 4 neutropenia will only be considered a DLT if it lasts longer than 7 days despite appropriate supportive care. Grade 4 thrombocytopenia will only be considered a DLT if it lasts longer than 7 days or is associated with greater then or equal to grade 3 bleeding event
Time Frame: 28 days
Measure: Number; unit: participants with DLT
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4
Number analyzed (Participants) | 3 | 3 | 6 | 6
participants with DLT | 0 | 0 | 1 | 1

2. Primary Outcome: Progression Free Survival (PFS) (Phase II)
Description: progression-free survival (PFS), defined as the time from randomization to the date the International Myeloma Working Group (IMWG) criteria for disease progression is met. If a patient initiates another anti-cancer treatment prior to disease progression, they will be censored at the date of initiation of this treatment. Patients will be randomized to treatment using the Pocock-Simon algorithm balancing the distribution of the following stratification factors between the two treatment arms: 1) ISS 1-2 disease vs. ISS 3 disease (current ISS stage based off screening beta 2 microglobulin and albumin) 2) High risk cytogenetics features: yes vs. no High risk cytogenetics features include: del(1p), gain of 1q, t(4;14), t(14;16), t(14; 20), del(17p) 3) Prior treatment with a proteasome inhibitor: yes vs. no
Time Frame: 3 years
Population: All eligible phase 2 patients were included in this analysis
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase II Arm I (Pomalidomide, Dexamethasone) | Phase II Arm II (Pomalidomide, Dexamethasone, Ixazomib)
Number analyzed (Participants) | 39 | 38
days | 228 [149 to 466] | 619 [245 to NA] — Upper limit not reached due to lack of events

3. Secondary Outcome: Incidence and Type of Dose Limiting Toxicities (DLTs) Graded According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (Phase I)
Description: These events are reported in the adverse events section of this report.
Time Frame: 44.5 months
Population: All enrolled phase 1 patients that were eligible and treated per protocol were evaluated for dose limiting toxicities. This excludes two dose level 2 patients, one dose level 3 patient and 5 dose level 4 patients.
Measure: Number; unit: participants with DLT
Groups:
- Phase 1 Dose Level 3: A 3 + 3 phase I dose escalation design was used to examine the safety profile and establish the MTD of IXA when given in combination with POM-DEX. Protocol therapy was administered over a 28-day cycle. IXA was given at a dose of 2.3 up to 4 mg by mouth on days 1, 8, and 15; POM at 2 up to 4 mg daily by mouth on days 1-21; and DEX 20 mg (age > 75 years) or 40 mg (age ≤ 75) by mouth on days 1, 8, 15, and 22 (Table 1). A new cycle of treatment was not to begin until the ANC was ≥ 1.0 × 109/L, platelets ≥ 50 × 109/L, and all other adverse events (AEs) had improved to grade 1 or baseline. Treatment continued until PD, the emergence of unacceptable toxicity, or patient request to discontinue protocol treatment. Dose Level 1 was 4mg POM-DEX and 3mg IXA.
- Phase 1 Dose Level 4: A 3 + 3 phase I dose escalation design was used to examine the safety profile and establish the MTD of IXA when given in combination with POM-DEX. Protocol therapy was administered over a 28-day cycle. IXA was given at a dose of 2.3 up to 4 mg by mouth on days 1, 8, and 15; POM at 2 up to 4 mg daily by mouth on days 1-21; and DEX 20 mg (age > 75 years) or 40 mg (age ≤ 75) by mouth on days 1, 8, 15, and 22 (Table 1). A new cycle of treatment was not to begin until the ANC was ≥ 1.0 × 109/L, platelets ≥ 50 × 109/L, and all other adverse events (AEs) had improved to grade 1 or baseline. Treatment continued until PD, the emergence of unacceptable toxicity, or patient request to discontinue protocol treatment. Dose Level 1 was 4mg POM-DEX and 4mg IXA.
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4
Number analyzed (Participants) | 3 | 3 | 6 | 6
participants with DLT | 0 | 0 | 1 | 1

4. Secondary Outcome: Incidence of Dose Reductions/Delays (Phase I)
Time Frame: 39 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4
Number analyzed (Participants) | 3 | 3 | 6 | 6
Participants | 2 | 3 | 6 | 5

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as partial response (PR), very good partial response (VGPR), complete response (CR), or stringent complete response (sCR) according to International Myeloma Working Group (IMWG) Uniform Response Criteria
Time Frame: 3 years
Population: All eligible and treated Phase II patients were included in analysis. Phase I patients were excluded from response analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Pomalidomide, Dexamethasone) | Arm II (Pomalidomide, Dexamethasone, Ixazomib)
Number analyzed (Participants) | 39 | 38
proportion of participants | .436 [.278 to .604] | .632 [.460 to .782]

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Disease response status is based on the IMWG criteria being held for two consecutive evaluations at least 4 weeks apart. Clinical benefit rate (CBR) is defined as proportion of patients with minimal response (MR) and better according to International Myeloma Working Group (IMWG) Uniform Response Criteria (Phase II)
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase II Arm I (Pomalidomide, Dexamethasone) | Phase II Arm II (Pomalidomide, Dexamethasone, Ixazomib)
Number analyzed (Participants) | 39 | 38
proportion of participants | .564 [.396 to .722] | .737 [.569 to .866]

7. Secondary Outcome: Disease Control Rate (DCR), Defined as Stable Disease (SD) and Better According to International Myeloma Working Group (IMWG) Uniform Response Criteria (Phase II)
Description: Proportion of patients that went two of more cycles of treatment without discontinuing treatment for progression or intolerability.
Time Frame: 42 days
Measure: Number (95% Confidence Interval); unit: proportion of partcipants
Arm/Group | Phase II Arm I (Pomalidomide, Dexamethasone) | Phase II Arm II (Pomalidomide, Dexamethasone, Ixazomib)
Number analyzed (Participants) | 39 | 38
proportion of partcipants | .949 [.827 to .994] | .921 [.786 to .983]

8. Secondary Outcome: Duration of Response (DOR), Calculated for All Patients Achieving an Objective Response, Partial Response (PR) or Better (Phase II)
Time Frame: Up to 3 years
Population: All eligible phase 2 responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II Arm I (Pomalidomide, Dexamethasone) | Phase II Arm II (Pomalidomide, Dexamethasone, Ixazomib)
Number analyzed (Participants) | 17 | 25
Months | 12.3 [2.8 to 37.0] | 23.7 [13.4 to 43.1]

9. Secondary Outcome: Overall Survival (OS) (Phase II)
Description: Overall survival was analyzed from the time of registration to the date of death or last known date living. Due to median OS time not being reached due to lack of deaths at the time of this report by either arm, the 2 year OS rate has been reported. This analysis censors living patients at 2 years.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: proportion of patients alive
Arm/Group | Phase II Arm I (Pomalidomide, Dexamethasone) | Phase II Arm II (Pomalidomide, Dexamethasone, Ixazomib)
Number analyzed (Participants) | 39 | 38
proportion of patients alive | .795 [.662 to .928] | .784 [.662 to .928]

10. Secondary Outcome: Time to Next Treatment (TNT) (Phase II)
Time Frame: Up to 3 years post-registration
Reporting Status: Not Posted, anticipated posting 2024-04

11. Secondary Outcome: Incidence, Type and Severity of Adverse Events, Graded According to National Cancer Institute (NCI) Common Terminology Criteria Adverse Events (CTCAE) Version 4.0 (Phase II)
Description: The count of paitents that experenced an adverse event is reported in this section. A full table of these events is reported in the adverse event section of this report.
Time Frame: 92 months
Measure: Count of Participants; unit: Participants
Groups:
- Phase II Arm II (Pomalidomide, Dexamethasone, Ixazomib) + Crossover Patients From Arm I: Patients receive pomalidomide, dexamethasone, and ixazomib as in Phase I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase II Arm I (Pomalidomide, Dexamethasone) | Phase II Arm II (Pomalidomide, Dexamethasone, Ixazomib) + Crossover Patients From Arm I | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4
Number analyzed (Participants) | 45 | 76 | 3 | 4 | 6 | 11
Participants | 22 | 33 | 2 | 2 | 4 | 6

12. Secondary Outcome: Response Rates (Overall Response Rate (ORR), Clinical Benefit Rate (CBR), Disease Control Rate (DCR) for All Patients on the Pomalidomide/Dexamethasone Arm at the Time of Cross-over to Pomalidomide/Dexamethasone/Ixazomib (Phase II)
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: proportion of partcipants
Groups:
- Arm I(Pomalidomide, Dexamethasone): Patients receive pomalidomide PO QD on days 1-21 and dexamethasone PO QD on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving disease progression may cross over to Arm II.
Arm/Group | Arm I(Pomalidomide, Dexamethasone)
Number analyzed (Participants) | 26
proportion of partcipants
  Overall Response Rate | .231 [.090 to .437]
  Clinical Benefit Rate | .269 [.116 to .478]
  Disease Control Rate | .962 [.804 to .999]

13. Secondary Outcome: Progression Free Survival (PFS) for All Patients on the Pomalidomide/Dexamethasone Arm at the Time of Cross-over to Pomalidomide/Dexamethasone/Ixazomib (Phase II)
Time Frame: Up to 3 years post-registration (at crossover)
Population: Arm 1 patients that chose to crossover to Arm 2 treatment (add IXA treatment).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Pomalidomide, Dexamethasone)
Number analyzed (Participants) | 26
months | 5.6 [3 to 12.9]

14. Secondary Outcome: Baseline Level of Perceived Fatigue and QOL, Assessed Using the Registration Fatigue/Uniscale Assessment Form (Phase II)
Description: Pre-treatment patient-report of fatigue and overall quality of life (based on a 10-point Likert scale). A higher number indicates a better quality of life where 10 is the best outcome and 0 is the worst.
Time Frame: baseline
Population: All patients that completed and returned the QoL survey
Measure: Number; unit: participants
Arm/Group | Arm I (Pomalidomide, Dexamethasone) | Arm II (Pomalidomide, Dexamethasone, Ixazomib)
Number analyzed (Participants) | 37 | 37
participants
  High QoL(7-10) | 21 | 27
  Medium or Low QoL (0-7) | 16 | 11

ADVERSE EVENTS:
Time Frame: 92 months
Description: All patients were included in mortality, only treated and evaluated patients are included in Adverse Events tables
Arm/Group | Phase II Arm I (Pomalidomide, Dexamethasone) | Phase II Arm II (Pomalidomide, Dexamethasone, Ixazomib) + Crossover Patients From Arm I | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4
All-Cause Mortality (participants affected / at risk) | 7/45 | 22/76 | 1/3 | 4/5 | 4/7 | 7/11
Serious Adverse Events (participants affected / at risk) | 22/45 | 33/76 | 2/3 | 2/4 | 4/6 | 6/11
Other Adverse Events (participants affected / at risk) | 45/45 | 76/76 | 3/3 | 4/4 | 6/6 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II Arm I (Pomalidomide, Dexamethasone) (N=45) | Phase II Arm II (Pomalidomide, Dexamethasone, Ixazomib) + Crossover Patients From Arm I (N=76) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level 2 (N=4) | Phase 1 Dose Level 3 (N=6) | Phase 1 Dose Level 4 (N=11)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve disease (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 3 (5) | 5 (7) | 1 (1) | 1 (1) | 0 (0) | 2 (4)
Lung infection (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (6) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II Arm I (Pomalidomide, Dexamethasone) (N=45) | Phase II Arm II (Pomalidomide, Dexamethasone, Ixazomib) + Crossover Patients From Arm I (N=76) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level 2 (N=4) | Phase 1 Dose Level 3 (N=6) | Phase 1 Dose Level 4 (N=11)
Anemia (Blood and lymphatic system disorders) | 31 (187) | 56 (420) | 1 (3) | 4 (6) | 6 (53) | 10 (114)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 5 (25) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 6 (53) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (2) | 3 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 4 (12) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 8 (37) | 0 (0) | 0 (0) | 1 (25) | 2 (4)
Cataract (Eye disorders) | 1 (2) | 5 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (3) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 7 (35) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
Watering eyes (Eye disorders) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (15)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 12 (59) | 20 (129) | 1 (3) | 1 (7) | 1 (14) | 5 (29)
Diarrhea (Gastrointestinal disorders) | 24 (85) | 44 (364) | 2 (6) | 2 (7) | 2 (6) | 5 (28)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 4 (21) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (6) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (12) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (14) | 8 (26) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (2) | 5 (8) | 0 (0) | 0 (0) | 1 (1) | 3 (12)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (28) | 33 (173) | 2 (6) | 1 (2) | 3 (8) | 4 (26)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (9) | 19 (32) | 0 (0) | 1 (1) | 0 (0) | 4 (11)
Chills (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 8 (25) | 25 (185) | 2 (9) | 0 (0) | 2 (15) | 1 (2)
Edema trunk (General disorders) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 39 (241) | 66 (647) | 2 (35) | 3 (24) | 6 (59) | 10 (132)
Fever (General disorders) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (7)
Flu like symptoms (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gen disord and admin site conds-Oth spec (General disorders) | 18 (99) | 20 (106) | 2 (17) | 2 (2) | 1 (4) | 5 (28)
Localized edema (General disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (7) | 1 (2)
Malaise (General disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pain (General disorders) | 3 (8) | 15 (40) | 0 (0) | 1 (1) | 2 (11) | 5 (17)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gum infection (Infections and infestations) | 2 (6) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 5 (8) | 14 (30) | 1 (1) | 2 (3) | 1 (1) | 2 (6)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Skin infection (Infections and infestations) | 1 (1) | 5 (13) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 6 (10) | 10 (13) | 2 (6) | 1 (2) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 7 (54) | 1 (16) | 0 (0) | 1 (5) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 5 (6) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (29) | 12 (37) | 1 (1) | 0 (0) | 1 (2) | 1 (18)
Alkaline phosphatase increased (Investigations) | 4 (4) | 6 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (20) | 9 (32) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Blood bilirubin increased (Investigations) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 1 (2) | 1 (2)
Creatinine increased (Investigations) | 8 (16) | 17 (87) | 1 (1) | 1 (1) | 1 (1) | 3 (16)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (2)
Investigations - Other, specify (Investigations) | 4 (4) | 4 (5) | 1 (22) | 1 (1) | 1 (7) | 1 (2)
Lymphocyte count decreased (Investigations) | 24 (101) | 44 (279) | 2 (33) | 3 (23) | 4 (53) | 8 (13)
Neutrophil count decreased (Investigations) | 31 (181) | 55 (404) | 1 (30) | 2 (7) | 6 (50) | 8 (45)
Platelet count decreased (Investigations) | 18 (46) | 48 (211) | 1 (33) | 2 (4) | 6 (36) | 10 (97)
Weight gain (Investigations) | 7 (9) | 13 (59) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Weight loss (Investigations) | 2 (3) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 15 (65) | 40 (264) | 1 (21) | 3 (6) | 3 (37) | 4 (13)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 7 (16) | 1 (3) | 1 (2) | 1 (4) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 19 (81) | 42 (235) | 0 (0) | 1 (1) | 1 (1) | 4 (85)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6) | 8 (16) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (5) | 13 (29) | 0 (0) | 0 (0) | 1 (6) | 1 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 7 (10) | 17 (29) | 1 (3) | 0 (0) | 2 (2) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 10 (41) | 14 (56) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 11 (15) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (27) | 19 (52) | 0 (0) | 0 (0) | 2 (4) | 1 (19)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 10 (86) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (31) | 17 (74) | 0 (0) | 0 (0) | 0 (0) | 4 (63)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (36) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (11) | 8 (33) | 0 (0) | 1 (2) | 2 (3) | 2 (15)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (6) | 4 (24) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 5 (18) | 5 (24) | 0 (0) | 0 (0) | 1 (3) | 2 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (29) | 14 (79) | 0 (0) | 1 (1) | 0 (0) | 2 (28)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3 (7) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (12) | 8 (50) | 1 (15) | 2 (2) | 0 (0) | 2 (12)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 8 (18) | 14 (90) | 1 (1) | 0 (0) | 0 (0) | 3 (5)
Dysgeusia (Nervous system disorders) | 2 (4) | 4 (17) | 2 (20) | 1 (1) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 7 (18) | 12 (42) | 2 (30) | 0 (0) | 1 (4) | 2 (6)
Lethargy (Nervous system disorders) | 0 (0) | 3 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 4 (5)
Paresthesia (Nervous system disorders) | 2 (4) | 2 (18) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 31 (298) | 57 (559) | 1 (3) | 3 (24) | 5 (56) | 7 (24)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 6 (31) | 9 (33) | 2 (32) | 0 (0) | 2 (15) | 1 (10)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 5 (8) | 7 (44) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 10 (30) | 10 (38) | 2 (3) | 1 (17) | 0 (0) | 4 (5)
Confusion (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 4 (7) | 11 (44) | 1 (2) | 1 (4) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 18 (85) | 25 (204) | 2 (19) | 2 (29) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 4 (5) | 5 (45) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 4 (9) | 4 (9) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Restlessness (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 4 (7) | 3 (20) | 0 (0) | 0 (0) | 0 (0) | 1 (14)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 4 (5) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (14) | 1 (3) | 1 (1) | 1 (2) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (22) | 16 (92) | 0 (0) | 0 (0) | 3 (11) | 3 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (17) | 1 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7) | 0 (0) | 1 (3) | 1 (3) | 2 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (22) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (6) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (16) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (10) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (16) | 1 (1) | 1 (13) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (23) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (22) | 13 (31) | 1 (1) | 0 (0) | 2 (4) | 3 (5)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 2 (4) | 5 (10) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 2 (2) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 3 (26) | 3 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 4 (32) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 9 (36) | 16 (103) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Hypotension (Vascular disorders) | 0 (0) | 5 (17) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 3 (6) | 0 (0) | 0 (0) | 1 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT02004275/Prot_SAP_000.pdf